CLINICAL TRIAL: NCT00602589
Title: An Open-label, Randomized, 3-way Crossover Study to Evaluate the Bioequivalence of an Oral Suspension Formulation, an Oral Solution Formulation, and the Marketed Tablet Formulation of Levofloxacin in Healthy Subjects
Brief Title: A Study to Evaluate the Bioequivalence of an Oral Suspension Formulation, an Oral Solution Formulation, and the Marketed Tablet Formulation of Levofloxacin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR011395
Record Dates: First submitted 2008-01-07; First posted 2008-01-28 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: open-label; randomized; crossover; bioequivalence
MeSH Terms: interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin oral suspension; Levofloxacin oral solution; and Levofloxacin marketed tablet formulations

SUMMARY:
The primary objective of the study was to assess the bioequivalence of the oral suspension formulation, the oral solution formulation, and the marketed tablet formulation of levofloxacin, with the marketed tablet as the reference.

DETAILED DESCRIPTION:
In this single-dose study conducted at at single center, 3 oral formulations of levofloxacin (tablet, suspension, and solution) were assessed for their bioequivalence in healthy men and women aged 18 to 55 years old. Subjects were assigned different treatments based on chance; both the researcher and the study participant knew the treatment being administered. The study consisted of a screening period, 3 open-label treatment periods separated by washout periods of at least 4 days between doses, and a post-treatment period. Subjects received a single dose of all 3 study formulations, administered as a single dose of each formulation on Day 1 of each treatment period. Blood samples were collected on Days 1, 2, and 3 of each treatment period immediately before dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 10, 14, 24, 30, 36, and 48 hours after dosing for measurement of levofloxacin concentration. Subjects were admitted to the study site prior to dosing and remained through the 48-hour measurements on Day 3. The post-treatment period included physical examination and clinical laboratory testing to ensure subject safety before being discharged from the study. Safety evaluations, including adverse event monitoring, standard clinical laboratory evaluations (hematology, serum chemistry, and urinalysis), vital sign monitoring, and physical examinations, were monitored throughout the study.

Two cohorts of 36 subjects each were enrolled in the study. The first cohort received a single dose of study drug and completed Period 1; the study was then stopped and reinitiated. Subjects from the first cohort completed early termination procedures; their data were included in safety analyses, however, no blood samples for levofloxacin concentrations were analyzed or included in pharmacokinetic analysis. Thirty-four subjects in the second cohort completed all study procedures. Levofloxacin oral suspension (125 mg/5 mL), levofloxacin oral solution (125 mg/5 mL), and levofloxacin tablet (500 mg) administered on Day 1 of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 18 to 55 years
* BMI between 18 and 30 kg/m2
* No prescription or over-the-counter medications for previous 14 days
* Negative tests for drug and alcohol abuse, HIV, hepatitis B and hepatitis C
* and Healthy based on medical history, physical examination, 12-lead electrocardiograms, toxicology, antigen, and antibody screens, and clinical laboratory evaluations

Exclusion Criteria:

* Allergic reaction to quinolones
* Clinically significant ECG or clinical laboratory abnormalities
* Creatinine clearance <=80 mL/min
* Acute illness within 7 days
* Nicotine use within 1 year
* Receipt of experimental drug or device within 60 days
* Pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2002-10; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the bioequivalence of the oral suspension formulation, the oral solution formulation, and the marketed tablet formulation of levofloxacin, on Days 1, 2, and 3, using the marketed tablet as the reference.

SECONDARY OUTCOMES:
Assessment of the bioequivalence of the oral suspension and solution formulations, on Days 1, 2, and 3, using the suspension formulation as the reference.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Click here to view the journal abstract from the study manuscript. — http://download.veritasmedicine.com/PDF/CR005824_alimentarypharmacologyandtherapeutics.pdf
- See also: An open-label, randomized, 3-way crossover study to evaluate the bioequivalence of an oral suspension formulation, an oral solution formulation, and the marketed tablet formulation of Levofloxacin in healthy subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=730&filename=CR011395_CSR.pdf